CLINICAL TRIAL: NCT05291130
Title: Evaluation Effectiveness of the Aesculap® Plasmafit Cementless Acetabular System in Combination With Vitelene® Polyethylene and Vitamin E Insert for Hip Arthroplasty
Brief Title: AESCULAP® Plasmafit® Cementless Acetabular System With Vitelene® Vitamin E Stabilized Highly Crosslinked Polyethylene
Status: Completed | Type: Observational
Sponsor: Federal State Budgetary Organization, Federal Center for Traumatology, Orthopedics and Arthroplasty (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-3
Record Dates: First submitted 2021-12-15; First posted 2022-03-22 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2022-03

CONDITIONS: Osteoarthritis, Hip; Rheumatic Arthritis; Degenerative Osteoarthritis
Keywords: Osteoarthritis hip; Orthopaedic surgery; Vitamin E crosslinked polyethylene; Hip arthroplasty; Ceramic femoral heads; Metal femoral heads
MeSH Terms: conditions — Osteoarthritis, Hip; Rheumatic Fever; Joint Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Plasmafit® Vitelene® Vitamin E ceramic femoral heads: Plasmafit® Acetabular Cup System with Vitelene® is a highly crosslinked polyethylene stabilized with vitamin E and bioceramic femoral heads
  Interventions: Device: Plasmafit® Vitelene® Vitamin E
- Plasmafit® Vitelene® Vitamin E metal femoral heads: Plasmafit® Acetabular Cup System with Vitelene® is a highly crosslinked polyethylene stabilized with vitamin E and metal femoral heads
  Interventions: Device: Plasmafit® Vitelene® Vitamin E
- Plasmafit® polyethylene metal femoral heads: Plasmafit® Acetabular Cup System with polyethylene and metal femoral heads

INTERVENTIONS:
Device: Plasmafit® Vitelene® Vitamin E — Plasmafit® Acetabular Cup System with an insert Aesculap ® Vitelene ® Vitamin E Stabilized Highly Crosslinked Polyethylene and BIOLOX delta Ceramic Femoral Head or ISODUR® Metal Femoral Heads
  Other Names: Plasmafit® Acetabular Cup System; BIOLOX delta Ceramic Femoral Head; ISODUR® Metal Femoral Heads
  Groups: Plasmafit® Vitelene® Vitamin E ceramic femoral heads; Plasmafit® Vitelene® Vitamin E metal femoral heads

SUMMARY:
Objectives of this study is evaluate effectivness of AESCULAP® Plasmafit® Plasmafit Cementless Acetabular System With Vitelene® Vitamin E Stabilized Highly Crosslinked Polyethylene compare to the sane sistem without Vitamin E, and ceramic or metal femoral heads

DETAILED DESCRIPTION:
Osteoarthritis is one most common disease in aged population, that most advanced stage needs surgical treatment. Surgical treatment usually include installation of implants. Every year new types of implants were fabricated from the new material. The effectiveness of this new devices need carefully independent assess in clinic.

ELIGIBILITY:
Inclusion Criteria:

* All patients who needs total knee replacement surgery
* Informed consent from the patients.

Exclusion Criteria:

-

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who need total knee replacmet surgury with a diagnosis
  * Pertrochanteric fracture
  * Disorder of continuity of tibia bone
  * Osteoarthritis of hip
  * Polyosteoarthritis
  * Acquired deformity of musculoskeletal system
  * Ankylosis of joint
  * Rheumatoid arthritis
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Functional assessments of hip joint replacement over time with Harris Hip Score (HHS) | 3 year follow-up
  The HHS is a measure of dysfunction of the hip joint. Consist of 10 items in 3 sections. Score <70 = poor result; 70-80 = fair, 80-90 = good, and 90-100 = excellent.
Functional assessments of knee joint replacement over time with Knee Society Score (KSS) | 3 year follow-up
  The KSS is a measure of dysfunction of the knee joint. The KSS has a two sections: "Knee Score" section (7 items) and a "Functional Score" section (3 items). Results can be interpreted with the following: 80-100 = excellent; score 70-79 = good; score 60-69 = fair; score <60 = poor.
Forgotten Joint Score-12 (FJS-12) for knee joint, modified Rankin scale | 3 year follow-up
  FJS-12 shows how much did the patient forget their artificial joint. Consists of 12 items, each item is answered within a 5-point Likert scale, as follows: 0: never (0 p); almost never (1 p); seldom (2 p); sometimes (3 p); and mostly (4 p). The initial raw data were converted to a scale ranging from 0 to 100 (worst to best).
Measuring postoperative pain using the visual analog scale for pain (VAS-P) | 3 year follow-up
  To measure pain intensity after surgery the patients choose the score on the 10 cm line scale with (VAS-P) rage from 0 ('no pain') to 10 (severe pain).
The modified Rankin scale (mRS) | 3 year follow-up
  mRS was used scale for measuring the degree of disability or dependence in the daily activities after joint replacement, with the following response options: 0: No symptoms at all; 1: No significant disability despite symptoms; able to carry out all usual duties and activities; 2: Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance; 3: Moderate disability; requiring some help, but able to walk without assistance; 4: Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance; 5: Severe disability; bedridden, incontinent and requiring constant nursing care and attention; 6: Dead

SECONDARY OUTCOMES:
The assessment of the assessment of quality of life | 3 year follow-up
  The assessment of quality of life using EQ-5D measure: mobility, self-care, usual activities, pain/discomfort and anxiety/depression based on a three-level version included "no problems, slight problems, moderate problems, severe problems, and unable to do/extreme".
Rentgenological assessments knee and hip replacement over time | 3 year follow-up
  Rentgenological results based on standing anteroposterior pelvic radiograph with assesment version, acetabular interclination, depth, height, stability of endoprosthesis components, signs of wear on the insert, presence of osteolysis zones. Installing additional locking screws, acetabular cup anteversion and inclination, limb length discrepancy after surgery.
Postoperative complications | 3 year follow-up
  Period of occurrence and type of complications are recorded
Revision surgery | 1 year follow-up
  The incidence of revision, time interval and types of incidence - one or two steps
The quality-adjusted life-year | 3 year follow-up
  Measure of the value of health outcomes with using the Short Form 36 (SF-36) health survey

CONTACTS AND LOCATIONS:
Overall Officials: Nikolai U Nikolaev, MD PhD, Study Chair — Federal State Budgetary Organization, Federal Center for Traumatology, Orthopedics and Arthroplasty
Locations (1):
- Federal Center for Traumatology, Orthopedics and Endoprosthetics, Cheboksary, Chuvashskaya Respublika, Russia